CLINICAL TRIAL: NCT00485459
Title: Efficacy, Tolerability, and Safety of Once-Daily Atomoxetine Hydrochloride Versus Placebo in Taiwanese Children and Adolescents With Attention-Deficit/Hyperactivity Disorder
Brief Title: Atomoxetine Hydrochloride Versus Placebo in Taiwanese Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8160; B4Z-TW-S010
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride
Drug: Placebo

SUMMARY:
The purpose of this protocol is to investigate the acute treatment efficacy, safety, and tolerability of atomoxetine on a once-daily dosing strategy in Taiwanese children and adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have ADHD that meet DSM-IV disease diagnostic criteria as well as severity criteria
* Subjects must be aged 6 to 16 years
* Subjects must not have taken any medication used to treat ADHD or they must have completed the washout procedures
* Subjects must be able to swallow capsules
* Subjects must be of normal intelligence in the judgment of the investigator. Normal intelligence is defined as being without evidence of significant general intellectual deficit and expected to achieve a score of 80 or more if formal IQ testing were administered.

Exclusion Criteria:

* Weigh less than 20 kg or more than 60 kg at study entry
* Have a history of Bipolar I or II disorder, psychosis, or pervasive developmental disorder
* Meet DSM-IV criteria for an anxiety disorder as assessed by the investigator
* Have a history of any seizure disorder (other than febrile seizures) or prior ECG abnormalities related to epilepsy, or subjects who have taken (or are currently taking) anticonvulsants for seizure control
* Subjects who have a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2004-02; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Test the hypothesis that atomoxetine administered as a single-daily dose provides superior efficacy compared with placebo in Taiwanese children and adolescents with ADHD

SECONDARY OUTCOMES:
Compare the improvement in symptoms associated with ADHD in children and adolescents achieved by once-daily dosing of atomoxetine or placebo
Compare the reduction in school-related symptoms between atomoxetine and placebo
Assess the safety and tolerability of once-daily dosing of atomoxetine

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Taipei, Taiwan

REFERENCES:
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com